CLINICAL TRIAL: NCT00723879
Title: Evaluation of Adherence Rate in Patients Receiving PegIntron / Rebetol (Weight Based) for Hepatitis C in Conjunction With a Patient Assistance Program.
Brief Title: Adherence in Patients Receiving PegIntron and Rebetol for Hepatitis C in Conjunction With a Patient Assistance Program (Study P04206)
Status: Terminated | Type: Observational
Why Stopped: Because of slow recruitment; Despite the study was started long time ago (Oct 2004), we have not reached the projected number of patients (150 patients)
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04206
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Hepatitis C, Chronic; Hepacivirus
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with hepatitis C: Patients receiving a patient assistance program during therapy for hepatitis C will be enrolled into this study. All patients will receive PegIntron plus Rebetol (according to the label) and the patient assistance program.
  Interventions: Biological: Peginterferon alfa-2b (SCH 54031); Drug: Ribavirin (SCH 18908); Behavioral: Patient assistance program

INTERVENTIONS:
Biological: Peginterferon alfa-2b (SCH 54031) — Peginterferon alfa-2b and ribavirin will be administered according to the products' labeling.
  Other Names: PegIntron
Drug: Ribavirin (SCH 18908) — Peginterferon alfa-2b and ribavirin will be administered according to the products' labeling.
  Other Names: Rebetol
Behavioral: Patient assistance program — Patient assistance programs will be classified as follows:
  1. medications, including psychiatric medications (antidepressants);
  2. other interventions, including nurse telephone calls and nurse support in the office: and
  3. educational literature about hepatitis C containing information about the disease, mode of transmission, complications, and treatment and treatment drawbacks that will be given to each patient at the start of treatment.

SUMMARY:
Patients receiving a patient assistance program during therapy for Hepatitis C will be enrolled into this study. All patients will receive PegIntron and Rebetol (according to the label) and the patient assistance program, which includes (1) medications used for treatment (psychiatric medications); (2) other interventions (nurse support); and (3) educational literature. This study will be compared to similar studies from other clinics using various patient support programs for the purpose of designing future comparative phase IV studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic hepatitis C naive to treatment

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving a patient assistance program during therapy for Hepatitis C will be enrolled into this study. All patients will receive PegIntron and Rebetol (according to the label) and the patient assistance program, which includes (1) medications used for treatment (psychiatric medications); (2) other interventions (nurse support); and (3) educational literature.
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2004-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who complete treatment with PegIntron plus Rebetol therapy for hepatitis C when administered with a patient assistance program. | NA (i.e. the study was terminated)
Average length of treatment for patients receiving a patient assistance program as part of their treatment for hepatitis C with PegIntron plus Rebetol. | NA (i.e. the study was terminated)